CLINICAL TRIAL: NCT06794671
Title: A Multicenter, Large-sample Case Registry Study to Evaluate Patient-reported Outcome and Medication Patterns With Vunakizumab for Inflammatory Skin Diseases
Brief Title: A Basket Trial of Vunakizumab in Inflammatory Skin Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0999
Record Dates: First submitted 2025-01-05; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Inflammatory Skin Diseases; Psoriasis
Keywords: inflammatory skin diseases; Psoriasis; vunakizumab
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a national multi-center, large sample size case registration clinical study. The registry population was patients with inflammatory skin diseases who were receiving treatment with vunakizumab. All outpatient and inpatient patients with inflammatory skin diseases who were receiving vunakizumab were eligible for enrollment. Patients' usual care was not affected by participation in the study. We only collected data in routine clinical practice.

The study had an enrollment period of 5 years or 10,000 patients were recruited early, whichever occurred first. All patients must provide written informed consent form before data collection, and each patient will be followed for 1 year to observe clinical progression.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ years；
* had adiagnosis of inflammatory skin disease；
* Is receiving or plans to receive vunakizumab for treatment;
* Patients provided written informed consent form.

Exclusion Criteria:

* no.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients woh had adiagnosis of inflammatory skin disease are receiving or plans to receive vunakizumab for treatment.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in DLQI scores over 52 weeks | Weeks 0 to 52
  DLQI: Dermatology Life Quality Index, range from 0 to 30, with higher scores indicating greater impact on quality of life

SECONDARY OUTCOMES:
Change from baseline in BSA over 52 weeks | Weeks 0 to 52
  BSA: body surface area
Change from baseline in IGA over 52 weeks | Weeks 0 to 52
  IGA: Investigator Global Assessment
Patterns of administration of vunakizumab for the treatment of different inflammatory skin diseases | Weeks 0 to 52
  The dose, interval, duration, and combined treatment of patients receiving vunakizumab were evaluated